CLINICAL TRIAL: NCT05137223
Title: The Development and Pilot Testing of a Caregiver-Child Shared Decision-Making Intervention to Improve Asthma in Urban Youth
Brief Title: BREATHE-Peds Pilot - I Focus Group Interviews
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Maureen George, Professor of Nursing, Columbia University Irving Medical Center, Columbia University
Other Study IDs: AAAT8015-I; 1R21NR019668-01A1 (NIH)
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2023-03

CONDITIONS: Asthma; Asthma in Children
Keywords: Asthma; Adolescents; Dyads; Shared decision-making; Minority health
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Adolescent Only Focus Groups: 20 early adolescents (ages 10-14) with physician-diagnosed persistent asthma (i.e., prescribed a controller medication) receiving care at a FQHC
- Caregiver Only Focus Groups: 20 informal caregivers (e.g., parent, grandparent) of early adolescents with physician-diagnosed persistent asthma receiving care at a FQHC
- Adolescent and Caregiver Focus Groups: 10 adolescents with physician-diagnosed persistent asthma receiving care at a FQHC and their caregivers (both of whom did not participate in either previous group for a total of 20 participants in the group cohort)

SUMMARY:
The overall aims of this study are to develop and pilot test BRief intervention to Evaluate Asthma THErapy (BREATHE)-Peds, a dyadic shared decision-making intervention, to improve asthma by supporting self-management among racial and ethnic minority early adolescents receiving care for uncontrolled asthma in federally-qualified health centers (FQHCs) in urban communities. Aim 1 (Phase I) involves developing the intervention through focus groups with early adolescents and caregivers. Aims 2 and 3 (Phase II) involve preliminary testing of the intervention through a pilot randomized controlled trial. This record is for Phase I only.

DETAILED DESCRIPTION:
Despite high asthma prevalence and morbidity among adolescents (highest among Black and Hispanic youth and early adolescents aged 10-14), there is a lack of developmentally appropriate interventions for this at-risk group. Racial and ethnic minority early adolescents have sub-optimal asthma self-management. Critical health behaviors that emerge during early adolescence affect lifelong patterns; therefore, early adolescence offers a unique opportunity to intervene. Additionally, successful self-management requires the right division of responsibility between adolescents and their caregivers. Thus, intervening simultaneously with early adolescents and their caregivers who can help support the adolescent's growing autonomy to self-manage their condition has the potential for a synergistic effect.

Prior studies have demonstrated the effects of improved asthma control of BREATHE, a brief one-time shared decision-making intervention for Black adults with uncontrolled asthma that utilizes motivational interviewing delivered by primary care providers. This study (i.e., Phase I) attempts to build on these promising results by adapting BREATHE to caregiver-early adolescent dyads. Phase I of the study will involve conducting up to 6 focus groups to identify components of BREATHE that are relevant to racial and ethnic minority early adolescents with uncontrolled asthma receiving care at FQHCs in urban communities and their caregivers. Focus groups will be composed of ~10 participants each: (a) two groups of early adolescents aged 10-14 with asthma; (b) two groups of the caregivers of the youth in Group A; and (c) two groups of adolescent-caregiver dyads who did not participate in Group A or B. Investigators will use the focus group results to write BREATHE-Peds, making modifications based on feedback from two primary care providers and two pediatric pulmonologists.

ELIGIBILITY:
Inclusion Criteria (adolescents):

* Aged 10-14 years
* Physician-diagnosed persistent asthma (defined as being prescribed a controller medication)

Exclusion Criteria (adolescents):

* Serious mental health conditions
* Developmental delay

Inclusion Criteria (caregivers):

* Informal caregivers (e.g., parent, grandparent) of adolescents aged 10-14 years with physician-diagnosed persistent asthma

Exclusion Criteria (caregivers):

* Serious mental health conditions

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Early adolescents (aged 10-14 years) with persistent uncontrolled asthma receiving care in federally-qualified health centers and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Number of participants who successfully complete the focus group | up to 12 months
  Focus groups will be held with early adolescents and caregivers to identify relevant components of a pre-existing intervention (i.e., BREATHE) for a new intervention (i.e., BREATHE-Peds). Information collected during these focus groups will aid in the design/implementation of the intervention to be pilot-tested in Phase II.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen George, PhD, Principal Investigator — Columbia University; Jean-Marie Bruzzese, PhD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Urban Health Plan: Adolescent Health and Wellness, The Bronx, New York
  - Urban Health Plan: El Nuevo San Juan, The Bronx, New York
  - Urban Health Plan: Bella Vista, The Bronx, New York

REFERENCES:
- [Background] Centers for Disease Control. Asthma Surveillance Data. Retrieved from https://www.cdc.gov/asthma/asthmadata.htm October 20, 2020.
- [Background] Zahran HS, Bailey CM, Damon SA, Garbe PL, Breysse PN. Vital Signs: Asthma in Children - United States, 2001-2016. MMWR Morb Mortal Wkly Rep. 2018 Feb 9;67(5):149-155. doi: 10.15585/mmwr.mm6705e1. PMID 29420459
- [Background] Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007. Pediatrics. 2009 Mar;123 Suppl 3:S131-45. doi: 10.1542/peds.2008-2233C. PMID 19221156
- [Background] Claudio L, Stingone JA, Godbold J. Prevalence of childhood asthma in urban communities: the impact of ethnicity and income. Ann Epidemiol. 2006 May;16(5):332-40. doi: 10.1016/j.annepidem.2005.06.046. Epub 2005 Oct 20. PMID 16242960
- [Background] Lara M, Akinbami L, Flores G, Morgenstern H. Heterogeneity of childhood asthma among Hispanic children: Puerto Rican children bear a disproportionate burden. Pediatrics. 2006 Jan;117(1):43-53. doi: 10.1542/peds.2004-1714. PMID 16396859
- [Background] Bruzzese JM, Bonner S, Vincent EJ, Sheares BJ, Mellins RB, Levison MJ, Wiesemann S, Du Y, Zimmerman BJ, Evans D. Asthma education: the adolescent experience. Patient Educ Couns. 2004 Dec;55(3):396-406. doi: 10.1016/j.pec.2003.04.009. PMID 15582346
- [Background] Dahl RE, Allen NB, Wilbrecht L, Suleiman AB. Importance of investing in adolescence from a developmental science perspective. Nature. 2018 Feb 21;554(7693):441-450. doi: 10.1038/nature25770. PMID 29469094
- [Background] Williams PG, Holmbeck GN, Greenley RN. Adolescent health psychology. J Consult Clin Psychol. 2002 Jun;70(3):828-42. PMID 12090386
- [Background] Maggs JL, Schulenberg J, Hurrelmann K. Developmental transitions during adolescence: health promotion implications. In: Schulenberg J, Maggs JL, Hurrelman K, eds. Health Risks and Developmental Transitions During Adolescence. New York: Cambridge University Press. 1997;522-546.
- [Background] Klok T, Kaptein AA, Brand PLP. Non-adherence in children with asthma reviewed: The need for improvement of asthma care and medical education. Pediatr Allergy Immunol. 2015 May;26(3):197-205. doi: 10.1111/pai.12362. PMID 25704083
- [Background] Rhee H, Belyea MJ, Brasch J. Family support and asthma outcomes in adolescents: barriers to adherence as a mediator. J Adolesc Health. 2010 Nov;47(5):472-8. doi: 10.1016/j.jadohealth.2010.03.009. Epub 2010 May 14. PMID 20970082
- [Background] Yang TO, Sylva K, Lunt I. Parent support, peer support, and peer acceptance in healthy lifestyle for asthma management among early adolescents. J Spec Pediatr Nurs. 2010 Oct;15(4):272-81. doi: 10.1111/j.1744-6155.2010.00247.x. PMID 20880275
- [Background] Bruzzese JM, Stepney C, Fiorino EK, Bornstein L, Wang J, Petkova E, Evans D. Asthma self-management is sub-optimal in urban Hispanic and African American/black early adolescents with uncontrolled persistent asthma. J Asthma. 2012 Feb;49(1):90-7. doi: 10.3109/02770903.2011.637595. Epub 2011 Dec 7. PMID 22149141
- [Background] Holley S, Morris R, Knibb R, Latter S, Liossi C, Mitchell F, Roberts G. Barriers and facilitators to asthma self-management in adolescents: A systematic review of qualitative and quantitative studies. Pediatr Pulmonol. 2017 Apr;52(4):430-442. doi: 10.1002/ppul.23556. Epub 2016 Oct 7. PMID 27717193
- [Background] Bruzzese JM, Unikel L, Gallagher R, Evans D, Colland V. Feasibility and impact of a school-based intervention for families of urban adolescents with asthma: results from a randomized pilot trial. Fam Process. 2008 Mar;47(1):95-113. doi: 10.1111/j.1545-5300.2008.00241.x. PMID 18411832
- [Background] George M, Bruzzese JM, Lynn S Sommers M, Pantalon MV, Jia H, Rhodes J, Norful AA, Chung A, Chittams J, Coleman D, Glanz K. Group-randomized trial of tailored brief shared decision-making to improve asthma control in urban black adults. J Adv Nurs. 2021 Mar;77(3):1501-1517. doi: 10.1111/jan.14646. Epub 2020 Nov 29. PMID 33249632